CLINICAL TRIAL: NCT02019238
Title: Second Randomization Study to Assess Efficacy of Different Ablation Strategies in Achieving Long-Term Arrhythmia Control in Patients With Persistent or Long Standing Persistent Atrial Fibrillation: RASTA XT Study
Brief Title: Second Study to Assess Different Ablation Strategies in Achieving Long-Term Arrhythmia Control in Patients With Persistent or Long Standing Persistent Atrial Fibrillation
Acronym: RASTA XT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI discretion
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 818358; 818358 (Other: University of Penn sylvania)
Record Dates: First submitted 2013-10-30; First posted 2013-12-24 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1-Standard PVI ablation (Placebo Comparator): Pulmonary Vein Isolation procedure combined with ablation of documented non-PV triggers of AF
  Interventions: Other: Pulmonary Vein Isolation procedure
- Group 2-PVI with empiric ablation (Active Comparator): Pulmonary Vein Isolation procedure combined with empiric ablation of common sites of non-PV triggers of AF and locations that may sustain AF sources on long term arrhythmia control
  Interventions: Other: Pulmonary Vein Isolation procedure

INTERVENTIONS:
Other: Pulmonary Vein Isolation procedure — comparing the efficacy of PVI ablation vs PVI combined with empiric ablation
  Other Names: PVI ablation procedure

SUMMARY:
Pulmonary vein isolation (PVI) combined with empiric ablation of either common sites of non-PV triggers of Atrial Fibrillation (AF) and locations that may sustain stable AF sources should be more efficacious than PVI combined with ablation of only documented non-PV triggers of AF in achieving long-term arrhythmia control in patients with persistent or long standing persistent AF.

DETAILED DESCRIPTION:
The AF ablation procedure has evolved considerably and currently the most accepted technique involves creation of circumferential Radiofrequency Ablation lesions around PV ostia (encircling wide areas around the left and right sided veins). We have found that targeting areas outside the pulmonary veins that trigger atrial premature beats of AF is important for optimizing the success of AF ablation. The methodology of additional lesion creation remains non-uniform, lacks mechanistic insights, and there is paucity of prospective randomized comparison on the long term efficacy and safety of various lesion combinations in achieving AF control. Our group recently conducted randomized study (RASTA Trial) that compared PVI combined with ablation of documented non-PV triggers (standard AF ablation strategy) of AF to two other strategies i.e. 1. PVI combined with empiric ablation at common non-PV trigger sites of AF, 2. PVI combined with ablation of locations demonstrating complex fractionated electrograms. In this study comprising 156 subjects with persistent and/or long standing persistent AF, the investigators found that the standard AF ablation strategy was as efficacious as PVI combined with empiric ablation at common non-PV trigger sites of AF and both of these approaches were significantly better than PVI combined with ablation of locations demonstrating complex fractionated electrograms. Our study also showed that when compared to the standard AF ablation strategy (PVI combined with ablation of documented non PV AF triggers), PVI combined with empiric ablation at common locations of AF triggers in the left and right atria showed 22% higher odds of achieving freedom from atrial arrhythmias and 33% higher odds of achieving arrhythmia control at one year. Although this difference may have been clinically meaningful, it did not reach statistical significance because this study was powered to test for a difference of ≥30% between groups. Thus, in the current proposal the investigators hope to show statistical difference in the outcomes between these two strategies by increasing the sample size which will provide adequate power to show a 20% difference in the primary outcome. Also, the investigators hope to enhance the outcome in the study arm (PVI combined with empiric ablation at common locations of AF triggers) by also targeting empirically locations in the left and right atria that have been shown in recent studies to be focal sources and rotors that maintain AF.

ELIGIBILITY:
Inclusion Criteria:

* All patients of age ≥ 18 years, undergoing their first ablation procedure that meet American College of Cardiology / American Heart Association defined criteria for persistent or long standing persistent AF will be eligible to participate in the proposed study. This includes patients with a history of AF episodes lasting at least 7 days and requiring at least 2 cardioversions.

Exclusion Criteria:

* Patients with paroxysmal AF (self-terminating episodes lasting < 7 day)
* Patients who have had a previous AF ablation procedure
* Failure to obtain informed consent
* Patients < 18 years of age. Investigators will plan to exclude paroxysmal AF patients and concentrate on patients with persistent or long standing persistent AF who may require further ablation to achieve better outcomes. Patients who have undergone previous AF ablation procedure will be excluded since the prior methodology used may confound the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Primary | 1 year
  Compare PVI strategies in group 1 (documented non-PV triggers of AF) to group 2 (PVI combined with empiric ablation of common sites) over 12 months to assess for recurrence of atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Dixit, MD, Principal Investigator — University of Pensylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States